CLINICAL TRIAL: NCT04959526
Title: Comparison of Shear-wave Elastography to State-of-the-art Respiratory Function Testing to Measure the Range of Forces Generated by the Diaphragm Muscle
Brief Title: Shear-wave Elastography Compared to Respiratory Function Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carlos B Mantilla, MD, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-003003
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Function Loss; Respiratory Complication
Keywords: Elastography; Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Respiratory Function Testing (Experimental): All subjects will receive standard respiratory function testing and ultrasound-based elastography measurements across various behaviors and conditions
  Interventions: Diagnostic Test: Shear-wave elastography

INTERVENTIONS:
Diagnostic Test: Shear-wave elastography — Ultrasound based imaging of diaphragm muscle activity

SUMMARY:
The purpose of this study is to evaluate the relationship between transdiaphragmatic pressure (Pdi) and diaphragm shear-wave elastography (SWE) during state-of-the-art respiratory muscle testing including volitional efforts (e.g., maximal inspiratory pressure, maximal expiratory pressure, Valsalva maneuver), as well as maximal phrenic nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

- Adult male and female healthy volunteers.

Exclusion Criteria:

* Volunteers who are pregnant.
* Volunteers with known pulmonary pathology (COPD, asthma requiring routine treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Shear wave speed | 3 hours
  Elastography of the diaphragm muscle across various behaviors and conditions

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Matilla, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No